CLINICAL TRIAL: NCT02932189
Title: Use of a New Isokinetic Device Oriented by Software for Inspiratory Muscle Training in Prolonged Weaning
Brief Title: Use of a New Isokinetic Device for Inspiratory Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Jocemir Ronaldo Lugon, MD, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: isokinetic device
Record Dates: First submitted 2016-09-19; First posted 2016-10-13 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Respiration, Artificial
Keywords: Mechanical Ventilator Weaning; Respiratory Muscle Training; Mortality Rate
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Procedure: Ventilator weaning in the conventional way with a tracheal collar.
- Intervention (Experimental): Procedure: Ventilator weaning with a tracheal collar after inspiratory muscle training with an isokinetic device.
  Device: K5 Power Breath
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — For the inspiratory muscle training, an isokinetic device (K5 Power Breath, United Kingdom) will be attached to the artificial airway.
  Arms: Intervention

SUMMARY:
Introduction:

It is well established that physical fitness improves muscle performance either in sedentary people or in athletes. In this regard, specific exercises for respiratory muscles can result in better functional performance in hospitalized individuals, especially in critically ill patients in prolonged weaning.

Objectives:

To compare the following variables between intervention and control patients: success in weaning, free time off ventilator on ICU after weaning, and gain of muscle strength with the use of the inspiratory muscle training (IMT).

Patients and methods:

Prospective randomized controlled clinical trial. Only individuals on prolonged weaning will be enrolled. They will undergo IMT or will be managed in a conventional manner. The primary endpoint will be successful weaning. In addition, other variables such as free time off ventilator on ICU after weaning and muscle strength will be measured. In addition, mortality in the ICU, inside the hospital and after discharge will be followed for one year after study entrance.

Expected results:

According to the working hypothesis, it is expected that the performance of patients undergoing IMT will be superior to the conventional treatment. Also, their time to mortality is expected to be longer.

DETAILED DESCRIPTION:
The control group only performed inspiratory muscle training (IMT) with the use of the T-piece. From the first day of prolonged weaning, patients would remain in spontaneous breathing progressing their stay time each day, respecting the criteria already mentioned for interruption and return to mechanical ventilation in support pressure mode.

The intervention group, in addition to the protocol described above, would undergo inspiratory muscle training with the POWER breathe K-5 (UK) device. POWER breathe K-5 will be employed once a day, with an initial loading of 40% of maximal inspiratory strength in a schedule of 30 repetitions. This number of repetitions could be reached in one to 6 sessions depending on the respiratory muscle force of the patient. Most of the times more than one session were required. Typically, subjects performed two to six sessions of 5 to 15 breaths per day, with two minutes rest in ventilation pressure support mode. When the patient was unable to comply with the schedule, the training session was interrupted at a total of 3 minutes. The load was planned to be adjusted weekly with a 5 to 10% increase until 60% of the maximal inspiratory strength was reached with a total time of 10 minutes or 100 breaths. After training with POWER breathe K-5 (UK), the patient would return to mechanical ventilation in support pressure mode for 30-60 minutes, and then follow the conventional T-piece protocol. The IMT was conducted normally between 08h and 10h, Monday through Friday.

All study subjects would be under continuous surveillance through the multi-parameter DX 2010 monitor (Dixtal, São Paulo, SP, Brazil), which records the electrocardiogram, heart rate, peripheral oxygen saturation and systemic arterial pressure. At any sign of instability, the IMT was interrupted and the patient returned to the ventilatory support and/or supplemental oxygen therapy for recovery.

The trial was stopped if at least one of the following intolerance criteria was present: SaO2<90% or PaO2 <60 mm Hg with FIO2 >0.4; PaCO2 > 50 mm Hg or increased by > 8 mm Hg; arterial pH < 7.33 or decreased by 0.07 or more; breathing frequency > 35 breaths/min or increased by 50% for 5 min or longer; heart rate > 140 beats/min or a sustained increase or decrease of > 20%; mean blood pressure > 130 or < 70 mm Hg; or presence of agitation, diaphoresis, disorientation, or depressed mental status.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 18 on mechanical ventilation
* Able to initiate ventilator weaning.

Exclusion Criteria:

* Positive serology for HIV
* Other immunesupressive conditions
* Life expectancy less than 12 months
* Spinal cord injury above T8
* Mechanical ventilation started at another institution
* Body mass index >35 kg/m2.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Successful weaning | one year
  defined by 48 hours on spontaneous ventilation after ventilator withdrawal

SECONDARY OUTCOMES:
Change in maximal inspiratory strength in cm H2O as measured by the digital manovacuometer MVD300 for 60 seconds | one year
  Assessment of inspiratory strength by the maximal inspiratory pressure and the timed inspiratory effort index
Change in the timed inspiratory effort index in cm H2O/sec as calculated by the ratio of the maximal inspiratory pressure and time demanded to reach it as measured by the digital manovacuometer MVD300 for 60 seconds | one year
  Assessment of inspiratory strength by the maximal inspiratory pressure and the timed inspiratory effort index
Time off the ventilator in the ICU in days. | one year
  Assessment of the time the patients are kept in the ICU after the successful weaning,

OTHER OUTCOMES:
Mortality rate | two years
  mortality will be analysed for one year after entrance in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jocemir R Lugon, MD, PhD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Hospital Naval Marcilio Dias, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] da Silva Guimaraes B, de Souza LC, Cordeiro HF, Regis TL, Leite CA, Puga FP, Alvim SH, Lugon JR. Inspiratory Muscle Training With an Electronic Resistive Loading Device Improves Prolonged Weaning Outcomes in a Randomized Controlled Trial. Crit Care Med. 2021 Apr 1;49(4):589-597. doi: 10.1097/CCM.0000000000004787. PMID 33332819